CLINICAL TRIAL: NCT00293384
Title: Pilot Study Evaluating Aprepitant (MK-869) for Prevention of Nausea & Vomiting Secondary to High Dose Cyclophosphamide Administered to Patients Underging Undergoing Peripheral Hematopoietic Progenitor Cell Mobilization Prior to Autologous Transplantation
Brief Title: Aprepitant, Granisetron, & Dexamethasone in Preventing Nausea & Vomiting in Pts. Receiving Cyclophosphamide Before a Stem Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Muneer Abidi, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000456201; P30CA022453 (NIH); WSU-D-2797 (Other: Karmanos Cancer Institute); WSU-0504001728 (Other: Wayne State University - Human Investigation Committee)
Record Dates: First submitted 2006-02-16; First posted 2006-02-17 (Estimated); Results first posted 2014-10-03 (Estimated); Last update posted 2016-03-15 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Neoplasms; Nausea and Vomiting; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: nausea and vomiting; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); accelerated phase chronic myelogenous leukemia; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; atypical chronic myeloid leukemia, BCR-ABL negative; blastic phase chronic myelogenous leukemia; chronic eosinophilic leukemia; primary myelofibrosis; chronic myelomonocytic leukemia; chronic neutrophilic leukemia; chronic phase chronic myelogenous leukemia; de novo myelodysplastic syndromes; disseminated neuroblastoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; myelodysplastic/myeloproliferative neoplasm, unclassifiable; nodal marginal zone B-cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II small lymphocytic lymphoma; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent neuroblastoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; recurrent small lymphocytic lymphoma; recurrent malignant testicular germ cell tumor; refractory chronic lymphocytic leukemia; refractory hairy cell leukemia; refractory multiple myeloma; relapsing chronic myelogenous leukemia; secondary acute myeloid leukemia; secondary myelodysplastic syndromes; splenic marginal zone lymphoma; stage I multiple myeloma; stage II multiple myeloma; stage II ovarian epithelial cancer; stage III adult Burkitt lymphoma; stage III adult Hodgkin lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III chronic lymphocytic leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage III marginal zone lymphoma; stage III multiple myeloma; stage III ovarian epithelial cancer; stage III small lymphocytic lymphoma; stage III malignant testicular germ cell tumor; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV adult Burkitt lymphoma; stage IV adult Hodgkin lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV breast cancer; stage IV chronic lymphocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; stage IV marginal zone lymphoma; stage IV ovarian epithelial cancer; stage IV small lymphocytic lymphoma
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Nausea; Vomiting; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Congenital Abnormalities; Leukemia, Myeloid, Accelerated Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Myelomonocytic, Chronic; Leukemia, Neutrophilic, Chronic; Leukemia, Myeloid, Chronic-Phase; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Carcinoma, Ovarian Epithelial; Leukemia, Lymphocytic, Chronic, B-Cell; Testicular Neoplasms; Leukemia, Hairy Cell | interventions — Aprepitant; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; dexamethasone 21-phosphate; dexamethasone acetate; Granisetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Aprepitant, Dexamethasone, Cytoxan & Kytril (Experimental): Day 1: 1 mg of Kytril orally or I.V., 10 mg of Dexamethasone orally, and Aprepitant 125 mg orally, 1 hour prior to cyclophosphamide administration.
  Cyclophosphamide 4gm/m2 I.V. over 90 - 120 minutes.
  Days 2 & 3: Aprepitant 80 mg once daily in the morning.
  Interventions: Drug: Aprepitant; Drug: Cyclophosphamide; Drug: Dexamethasone; Drug: Granisetron hydrochloride

INTERVENTIONS:
Drug: Aprepitant — Aprepitant 80mg once daily in the morning on days 2 and 3
  Other Names: Emend
Drug: Cyclophosphamide — Cyclophosphamide 4 gm/m2 I.V. over 90-120 minutes
  Other Names: Cytoxan®; Neosar®
Drug: Dexamethasone — Dexamethasone orally 10 mg 1 hour prior to cyclophosphamide administration.
  Other Names: Decadron; Diodex; Hexadrol; Maxidex; Dexamethasone Sodium Phosphate; Dexamethasone Acetate
Drug: Granisetron hydrochloride — Kytril 1 mg orally or I.V., 1 hour prior to cyclophosphamide administration.
  Other Names: KYTRIL®

SUMMARY:
RATIONALE: Antiemetic drugs, such as aprepitant, granisetron, and dexamethasone, may help lessen or prevent nausea and vomiting in patients treated with chemotherapy.

PURPOSE: This clinical trial is studying how well giving aprepitant together with granisetron and dexamethasone works in preventing nausea and vomiting in patients receiving cyclophosphamide before undergoing an autologous stem cell transplant.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the efficacy of the addition of aprepitant in controlling acute vomiting with the standard prophylactic anti-emetic combination of granisetron hydrochloride and dexamethasone in patients receiving therapy comprising high-dose cyclophosphamide to mobilize stem cells prior to leukapheresis for autologous stem cell transplantation.

Secondary

* Evaluate the efficacy of the addition of aprepitant in controlling delayed vomiting in these patients.
* Evaluate the efficacy of the addition of aprepitant in controlling overall nausea in these patients.
* Identify side effects of the addition of aprepitant to this regimen in these patients.

OUTLINE: Patients receive granisetron hydrochloride orally or IV and oral dexamethasone, followed 1 hour later by cyclophosphamide IV over 2 hours on day 1. Patients also receive oral aprepitant once daily on days 1-3. Treatment continues in absence of unacceptable toxicity.

After completion of study treatment, patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing autologous peripheral blood stem cell transplantation and stem cell mobilization using cyclophosphamide
* Candidate (per institutional requirements) for autologous peripheral blood stem cell transplantation

  * No psychiatric illness or multi-system organ failure
* No nausea at baseline

PATIENT CHARACTERISTICS:

* SWOG performance status 0-2
* Fewer than 5 alcoholic drinks per day within the past year
* No current illness requiring chronic systemic steroids or requirement for chronic use of anti-emetics
* No gastrointestinal obstruction or active peptic ulcer disease
* AST and ALT ≤ 3 times upper limit of normal (ULN)
* Bilirubin ≤ 3 times ULN
* Alkaline phosphatase ≤ 3 times ULN
* Creatinine ≤ 2 mg/dL
* No known hypersensitivity to any component of the study regimen
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No unrelenting hiccups

PRIOR CONCURRENT THERAPY:

* No chronic therapeutic warfarin > 1 mg dose per day
* No other concurrent investigational agents
* No concurrent oral contraceptives (except for stopping menses), tolbutamide, phenytoin, midazolam, ketoconazole, rifampin, paroxetine hydrochloride, or diltiazem hydrochloride
* No concurrent illegal drugs

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-10; Primary Completion 2009-06 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muneer H. Abidi, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aprepitant, Dexamethasone, Cytoxan & Kytril: Day 1: 1 mg of Kytril orally or I.V., 10 mg of Dexamethasone orally, and Aprepitant 125 mg orally, 1 hour prior to cyclophosphamide administration.
  Cyclophosphamide 4gm/m2 I.V. over 90 - 120 minutes.
  Days 2 & 3: Aprepitant 80 mg once daily in the morning.
  Aprepitant: Aprepitant 80mg once daily in the morning on days 2 and 3
  Cyclophosphamide: Cyclophosphamide 4 gm/m2 I.V. over 90-120 minutes
  Dexamethasone: Dexamethasone orally 10 mg 1 hour prior to cyclophosphamide administration.
  Granisetron hydrochloride: Kytril 1 mg orally or I.V., 1 hour prior to cyclophosphamide administration.
Period: Overall Study
Arm/Group | Aprepitant, Dexamethasone, Cytoxan & Kytril
Started | 40
Completed | 35
Not Completed | 5
Not completed — Non-compliance | 2
Not completed — Missed dosage/study drug | 1
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Population: Patients who received all doses of the study drug were considered evaluable patients.
Arm/Group | Aprepitant, Dexamethasone, Cytoxan & Kytril
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Controlled Acute Vomiting
Description: No episodes of vomiting and no rescue medication during first 24 hours after cyclophosphamide administration.
Time Frame: at 0-24 hours
Population: Evaluable for response
Measure: Number; unit: participants
Arm/Group | Aprepitant, Dexamethasone, Cytoxan & Kytril
Number analyzed (Participants) | 35
participants | 20
Statistical Analysis 1: Comparison: Aprepitant, Dexamethasone, Cytoxan & Kytril; Optimal Simon design for phase II study. p0=45% p1=65%; Test type: Superiority or Other; p = 0.10, Simon optimal design — 85% statistical power; proportion = .57

2. Secondary Outcome: Delayed Vomiting Controlled
Time Frame: at 25-120 hours
Measure: Number; unit: participants
Arm/Group | Aprepitant, Dexamethasone, Cytoxan & Kytril
Number analyzed (Participants) | 35
participants | 22
Statistical Analysis 1: Comparison: Aprepitant, Dexamethasone, Cytoxan & Kytril; Test type: Superiority or Other; proportion = 0.63

3. Other Pre Specified Outcome: Overall Nausea Controlled
Time Frame: at 0-120 hours
Measure: Number; unit: participants
Arm/Group | Aprepitant, Dexamethasone, Cytoxan & Kytril
Number analyzed (Participants) | 35
participants | 31

4. Secondary Outcome: Toxicity Grade 3, 4, or 5
Time Frame: at 0-120 hours
Measure: Number; unit: participants
Arm/Group | Aprepitant, Dexamethasone, Cytoxan & Kytril
Number analyzed (Participants) | 35
participants | 2
Statistical Analysis 1: Comparison: Aprepitant, Dexamethasone, Cytoxan & Kytril; Test type: Superiority or Other; proportion = 0.06

ADVERSE EVENTS:
Arm/Group | Aprepitant, Dexamethasone, Cytoxan & Kytril
Serious Adverse Events (participants affected / at risk) | 10/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant, Dexamethasone, Cytoxan & Kytril (N=35)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1
Vomiting (Gastrointestinal disorders) | 2 (2)
Infection (Infections and infestations) | 2 (3)
Musculokeletal Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 6 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Mucositis (Metabolism and nutrition disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant, Dexamethasone, Cytoxan & Kytril (N=35)
Fever (General disorders) | 6 (6)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 24 (47)
Diarrhea (Gastrointestinal disorders) | 10 (12)
Vomiting (Gastrointestinal disorders) | 14 (16)
Infection (Infections and infestations) | 2 (2)
Headache (Nervous system disorders) | 7 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Tachycardia (Cardiac disorders) | 3 (3)
Neuropathy (Nervous system disorders) | 3 (3)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Hypokalemia (Metabolism and nutrition disorders) | 15 (19)
Pain- Cath site (General disorders) | 2 (2)
Fatigue (General disorders) | 17 (22)
Constipation (Gastrointestinal disorders) | 4 (4)
Belching (Gastrointestinal disorders) | 2 (2)
Lightheaded (Nervous system disorders) | 2 (2)
Acid Refulx (Gastrointestinal disorders) | 2 (2)
Weight gain (Investigations) | 2 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 3 (3)
Mucositis (Gastrointestinal disorders) | 2 (2)
Drowsy (Nervous system disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
There were no other significant limitations except for the details provided.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No